CLINICAL TRIAL: NCT03648671
Title: Spontaneous and Evoked Pain in Parkinson's Disease With Motor Fluctuations: an Observational, Prospective, Clinical and Neurophysiological Study in Patients Under L-dopa Add on Therapies.
Brief Title: Pain in Parkinson's Disease With Motor Fluctuations.
Acronym: PAINinPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Michele Tinazzi, MD, PhD, Full professor of Neurology, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 1470CESC
Record Dates: First submitted 2018-06-26; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease
Keywords: Safinamide; Pain; Parkinson
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PD with PAIN: 12 patients will undergo add-on drugs therapy with safinamide metansolfonato.
  Interventions: Drug: safinamide metansolfonato (12 weeks)
- PD without PAIN: 12 patients will undergo add-on drugs therapy with safinamide metansolfonato.
  Interventions: Drug: safinamide metansolfonato (12 weeks)
- PD with PAIN rasagilina: 12 patients will undergo add-on drugs therapy with rasagilina mesilato.
  Interventions: Drug: rasagilina mesilato (12 weeks)
- PD without PAIN rasagilina: 12 patients will undergo add-on drugs therapy with rasagilina mesilato.
  Interventions: Drug: rasagilina mesilato (12 weeks)

INTERVENTIONS:
Drug: safinamide metansolfonato (12 weeks) — safinamide metansolfonato
  Groups: PD with PAIN
Drug: safinamide metansolfonato (12 weeks) — safinamide metansolfonato
  Groups: PD without PAIN
Drug: rasagilina mesilato (12 weeks) — rasagilina mesilato
  Groups: PD with PAIN rasagilina
Drug: rasagilina mesilato (12 weeks) — rasagilina mesilato
  Groups: PD without PAIN rasagilina

SUMMARY:
Pain (spontaneous pain) is a fundamental non-motor symptom (NMS) of Parkinson's disease (PD) that is prevalent throughout the condition and often unrecognized and undertreated. The study of the scalp laser-evoked potentials (LEPs) (evoked pain) allows a non-invasive exploration of pain central pathways in humans. This technique proved useful in elucidating the physiopathology underlying different pain syndromes. This study has been conceived to study spontaneous pain (and/or evoked pain by laser stimulation) in PD patients (with or without pain) with motor fluctuations under drugs-on (Safinamide Metansolfonato or Rasagilina Mesilato).

DETAILED DESCRIPTION:
Pain (spontaneous pain) is a fundamental non-motor symptom (NMS) of Parkinson's disease (PD) that is prevalent throughout the condition and often unrecognized and undertreated. Different types of pain have been described in association with PD including musculoskeletal, dystonic, central and neuropathic pain. Although musculoskeletal pain is the most commonly reported, a number of patients experience multiple types of pain which are more frequent and disabling in the intermediate phase of disease and which ultimately have a significant negative impact on the patient's quality of life. Despite its relevance, the pathophysiological mechanisms underlying pain in PD are yet to be fully understood. An abnormal nociceptive input processing in the central nervous system leading to hypersensitivity to evoked pain probably underlies all the different pain types experienced by PD patients and also intervene in pain-free PD patients. Additional factors including female gender, depression, disease duration, motor complications, postural abnormalities, medical conditions associated with painful symptoms (osteoporosis, rheumatic or degenerative joint disease,) probably contribute to the quality and distribution of spontaneous pain. Abnormalities in pain processing may be the consequence of decreased basal ganglia dopaminergic neurotransmission, as dopamine has been demonstrated to modulate pain perception in supraspinal regions involved in the pain pathways, including insula, anterior cingulate cortex, thalamus and periaqueductal grey. Furthermore, a neurodegeneration involving non-dopaminergic systems (such as g-aminobutyric acid, glutamate, noradrenaline, and serotonin) that modulate pain processing in other regions of the central nervous systems may also play a relevant role. The variegated pain dimension experienced by PD patients makes its therapeutic management a demanding challenge for clinicians.

The study of the scalp laser-evoked potentials (LEPs) (evoked pain) allows a non-invasive exploration of pain central pathways in humans. This technique proved useful in elucidating the physiopathology underlying different pain syndromes. Some data show that LEPs are altered in PD, in both pain-free PD patients and in PD patients with different kinds of pain, with amplitude reduction in N2/P2 component. Acute levodopa challenge had no effect in normalizing the decreased pain threshold/LEPs observed in PD patients in early Parkinson's disease while in PD patients with motor complications it partially increased pain threshold. This is consistent with the hypothesis that motor complications and pain may share common pathophysiological mechanisms which include not only dopaminergic but also non-dopaminergic systems dysfunction (25).This study has been conceived to study spontaneous pain (and/or evoked pain by laser stimulation) in PD patients (with or without pain) with motor fluctuations under drugs-on (Safinamide Metansolfonato or Rasagilina Mesilato).

ELIGIBILITY:
Inclusion Criteria:

* PD patients with or without pain willing to participate in this study and able to sign the written informed consent
* To be included in the PD with pain group, the patient's intensity of pain must be moderate to severe over the last month, as reported by a numerical rating scores (NRS≥4) despite the optimal dopaminergic treatment
* No modification of dopaminergic drugs and analgesic therapy with FANS during the 28 days before starting the enrollment in this study.
* Diagnosis of idiopathic PD of ≥3 years duration
* Hoehn and Yahr stage I-III during OFF time
* Motor fluctuations (>1.5 hours' OFF time/day)
* Patients who would have been treated with add-on therapy irrespective to the present protocol

Exclusion Criteria:

* Patients under (or with previous assumptions) monoamine oxidase inhibitor therapy.
* Late-stage PD experiencing severe, disabling peak-dose or biphasic dyskinesia, or unpredictable or widely swinging symptom fluctuations
* "de novo" patients, patients in early stage or non-fluctuating patients
* Evidence of dementia (MMSE <24)
* Sign and symptoms suggestive of atypical parkinsonism
* Major psychiatric illnesses
* Severe and progressive medical illnesses
* Concomitant diseases potentially causing acute or chronic pain (i.e., rheumatologic conditions, severe polyneuropathy, and spine injuries)
* Treatments with tri-tetracyclic antidepressants, serotonin-norepinephrine reuptake inhibitors (SNRIs), opioids, neuroleptics, barbiturates and phenothiazines, pregabalin and gabapentin
* Any type of retinopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females patients with mid-to-late PD aged 30 to 80 years with or without chronic pain symptoms (duration >3 months) and motor fluctuations while receiving L-dopa alone or with other dopaminergic treatments.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Latency (ms) of N1/P1 complex. | Change from baseline at 12 weeks
  Laser-evoked potentials (LEPs) to explore the primary pain pathway will be assessed at each visit (V0 and V1). The technique of LEPs recording will be carried out as previously performed by our research group.
Latency (ms) of N2/P2 complex. | Change from baseline at 12 weeks
  Laser-evoked potentials (LEPs) to explore the primary pain pathway will be assessed at each visit (V0 and V1). The technique of LEPs recording will be carried out as previously performed by our research group.
Amplitude (microvolt) of N1/P1 complex. | Change from baseline at 12 weeks
  Laser-evoked potentials (LEPs) to explore the primary pain pathway will be assessed at each visit (V0 and V1). The technique of LEPs recording will be carried out as previously performed by our research group.
Amplitude (microvolt) of N2/P2 complex. | Change from baseline at 12 weeks
  Laser-evoked potentials (LEPs) to explore the primary pain pathway will be assessed at each visit (V0 and V1). The technique of LEPs recording will be carried out as previously performed by our research group.

SECONDARY OUTCOMES:
Body localization | Change from baseline at 12 weeks
  The presence of pain (yes/no, dichotomous variable) in one or more body parts: head, upper limbs, lower limbs, shoulders, neck, trunk , lumbar back, pelvis, knees.
King's Pain Scale for Parkinson's Disease | Change from baseline at 12 weeks
  (score)
Italian version of the brief pain inventory short form | Change from baseline at 12 weeks
  (score)
Clinical global impression of change | Change from baseline at 12 weeks
  (score)
The 39-Item Parkinson's Disease Questionnaire (PDQ-39) | Change from baseline at 12 weeks
  (score)
Numeric Rating Scale (NRS) | Change from baseline at 12 weeks
  (score)
Unified Parkinson's Disease Rating Scale | Change from baseline at 12 weeks
  (score)
Total daily off time | Change from baseline at 12 weeks
  Total daily off time will assessed by patient diaries reporting frequency and duration of the off periods (hours)
Off time following the first morning L-dopa dose | Change from baseline at 12 weeks
  (hours)
Age | One timepoint
  Age
Gender | One timepoint
  (male/female)
Schooling | One timepoint
  (years)
Job | One timepoint
  type of job
Weight | One timepoint
  (kg)
Disease duration | One timepoint
  (years)
Age at PD onset | One timepoint
  (years)
Laterality of PD symptom onset | One timepoint
  (right, left, bilateral)
Most Affected Side | One timepoint
  (right, left, bilateral)
Pain symptoms at PD onset | One timepoint
  (yes, no)
Dominant phenotype | One timepoint
  (Tremor, Bradikinetic/rigid, Mixed)
Modified H&Y | One timepoint
  (score)
Pharmacologic therapy for PD | One timepoint
  Pharmacologic therapy
Comorbilities | One timepoint
  Comorbilities
Mini-Mental State Examination | One timepoint
  (score)
Montreal Cognitive Assessment (MoCA) | One timepoint
  (score)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tinazzi, MD, PhD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Azienda ospedaliera universitaria integrata verona, Verona, Italy

REFERENCES:
- [Background] Defazio G, Berardelli A, Fabbrini G, Martino D, Fincati E, Fiaschi A, Moretto G, Abbruzzese G, Marchese R, Bonuccelli U, Del Dotto P, Barone P, De Vivo E, Albanese A, Antonini A, Canesi M, Lopiano L, Zibetti M, Nappi G, Martignoni E, Lamberti P, Tinazzi M. Pain as a nonmotor symptom of Parkinson disease: evidence from a case-control study. Arch Neurol. 2008 Sep;65(9):1191-4. doi: 10.1001/archneurol.2008.2. PMID 18779422
- [Background] Tinazzi M, Recchia S, Simonetto S, Tamburin S, Defazio G, Fiaschi A, Moretto G, Valeriani M. Muscular pain in Parkinson's disease and nociceptive processing assessed with CO2 laser-evoked potentials. Mov Disord. 2010 Jan 30;25(2):213-20. doi: 10.1002/mds.22932. PMID 20063386
- [Background] Tinazzi M, Recchia S, Simonetto S, Defazio G, Tamburin S, Moretto G, Fiaschi A, Miliucci R, Valeriani M. Hyperalgesia and laser evoked potentials alterations in hemiparkinson: evidence for an abnormal nociceptive processing. J Neurol Sci. 2009 Jan 15;276(1-2):153-8. doi: 10.1016/j.jns.2008.09.023. Epub 2008 Oct 26. PMID 18954878
- [Background] Tinazzi M, Del Vesco C, Defazio G, Fincati E, Smania N, Moretto G, Fiaschi A, Le Pera D, Valeriani M. Abnormal processing of the nociceptive input in Parkinson's disease: a study with CO2 laser evoked potentials. Pain. 2008 May;136(1-2):117-24. doi: 10.1016/j.pain.2007.06.022. Epub 2007 Aug 31. PMID 17765400
- [Background] Zambito-Marsala S, Erro R, Bacchin R, Fornasier A, Fabris F, Lo Cascio C, Ferracci F, Morgante F, Tinazzi M. Abnormal nociceptive processing occurs centrally and not peripherally in pain-free Parkinson disease patients: A study with laser-evoked potentials. Parkinsonism Relat Disord. 2017 Jan;34:43-48. doi: 10.1016/j.parkreldis.2016.10.019. Epub 2016 Oct 24. PMID 27836714